CLINICAL TRIAL: NCT00955253
Title: A Trial of Guanfacine, an Alpha 2 Adrenergic Agonist, for Spatial Neglect and Impaired Vigilance Following Stroke and Focal Brain Damage
Brief Title: Guanfacine for the Treatment of Spatial Neglect and Impaired Vigilance
Acronym: GASNIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO1234; NRES09/H0711/5 (Other: National Research Ethics Service); 2008-001160-36 (EudraCT Number)
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Stroke; Hemispatial Neglect
Keywords: Neglect; Attention; Vigilance; Stroke; Hemineglect; Unilateral Neglect; Spatial Neglect
MeSH Terms: conditions — Stroke; Perceptual Disorders | interventions — Guanfacine

STUDY DESIGN:
Intervention Model Description: Patients were tested on five consecutive days. On days 1, 3 and 5, they were tested on a task battery. On day 2, individuals received active drug or placebo, and on day 4 they received placebo if they had previously received active drug and vice versa. The order of administration of guanfacine and placebo was counterbalanced across patients, according to a pregenerated randomisation scheme. The clinician who administered the drugs and the tests was blind to the randomisation and the drug. The analyses presented here were performed by a different researcher, only after all data were collected. On both treatment days, patients were tested on the task battery twice: once immediately before guanfacine/placebo administration and once 2 hours after.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The order of administration of guanfacine and placebo was counterbalanced across patients, according to a pregenerated randomisation scheme. The clinician who administered the drugs and the tests was blind to the randomisation and the drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guanfacine (Day 2) then Placebo (Day 4) (Experimental): All patients received a single dose of guanfacine on Day 2 and a single dose of placebo on Day 4.
  Interventions: Drug: Guanfacine; Drug: Placebo
- Placebo (Day 2) then Guanfacine (Day 4) (Experimental): All patients received a single dose of placebo on Day 2 and a single dose of guanfacine on Day 4.
  Interventions: Drug: Guanfacine; Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine — 2mg oral guanfacine (encapsulated)
  Other Names: Estulic
Drug: Placebo — placebo

SUMMARY:
To find out if spatial neglect following stroke and brain injury can be reduced using guanfacine, a drug that was shown to improve neglect in two stroke patients in a previous pilot study (Malhotra et al, 2006). In this trial, the effects of guanfacine will be examined in a larger number of patients, and there will also be a systematic assessment of whether the drug is only effective in patients with particular patterns of brain damage.

DETAILED DESCRIPTION:
The current study has a double-blind crossover design where patients will receive a single 2mg dose of oral guanfacine and a single dose of placebo. They will receive one of these on Day 2 of the study period and the other on Day 4.

They will be tested daily on Days 1 to 5 so that any test repetition or long-term drug effects can be gauged.

On days 2 and 4 they will be tested twice-once prior to drug/placebo administration and again 90 minutes after drug/placebo administration.

Tests will include standard pen-and-paper tasks for neglect as well as computerised tests of sustained attention and visual exploration. In our published pilot study (Malhotra et al, 2006) there was a suggestion that patients without damage to frontal cortex were more likely to respond to guanfacine. In the current study we intend to test 10 patients with and 10 patients without frontal damage in order to test this further.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or more
* Greater than 2 weeks following stroke
* Ability to give consent
* Evidence of robust Visual Neglect when tested twice with cancellation tasks.

Exclusion Criteria:

* Less than 2 weeks following stroke
* Concomitant illness that may affect interpretation of any findings
* Labile blood pressure following stroke
* Systolic BP less than 100 mmHg and / or diastolic less than 70 mmHg
* New antihypertensive medication started within last 3 weeks
* Patients with hepatic or renal dysfunction
* Patients receiving other medications known to potentiate guanfacine's antihypertensive and hypotensive effects or cause torsade de pointes, specifically antipsychotics (including sultopride, chlorpromazine, thioridazine, amisulpiride, sulpiride, haloperidol), and moxifloxacin, baclofen, verapamil, quinidine, hydroquinidine, dispyramide, amiodarone, dofetilide, ibutilide, sotalol, pimozide, bepridil, cisapride, diphemanil, erythromycin IV, halofantrine, pentamidine, sparfloxacin, vincamine, alfuzosin, prazosin, terazosin, tamsulosin, amifostine
* Patients with diagnosis of brain tumour
* Patients with weight less than 55kg
* Patients who are pregnant
* Mothers who are breast feeding
* Patients with severe coronary insufficiency or myocardial infarction in previous 6 months
* Cognitive impairment, dysphasia or dementia that prevents patient from giving informed consent
* Severe mental impairment or physical handicap following stroke that prevents patients from giving consent or performing basic (standard clinical) tests for neglect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2014-03-28 (Actual); Study Completion 2014-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paresh A Malhotra, PhD MRCP, Principal Investigator — Imperial College London; Masud Husain, DPhil FRCP, Principal Investigator — University College, London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malhotra PA, Parton AD, Greenwood R, Husain M. Noradrenergic modulation of space exploration in visual neglect. Ann Neurol. 2006 Jan;59(1):186-90. doi: 10.1002/ana.20701. PMID 16261567
- [Result] Dalmaijer ES, Li KMS, Gorgoraptis N, Leff AP, Cohen DL, Parton AD, Husain M, Malhotra PA. Randomised, double-blind, placebo-controlled crossover study of single-dose guanfacine in unilateral neglect following stroke. J Neurol Neurosurg Psychiatry. 2018 Jun;89(6):593-598. doi: 10.1136/jnnp-2017-317338. Epub 2018 Feb 7. PMID 29436486

RESULTS

PARTICIPANT FLOW:
Groups:
- Guanfacine Then Placebo: This group individuals are randomised to receive Guanfacine at the first treatment session and Placebo at the second treatment session.
- Placebo Then Guanfacine: This group individuals are randomised to receive Placebo at the first treatment session and Guanfacine at the second treatment session.
Period: First Intervention (Day 2)
Arm/Group | Guanfacine Then Placebo | Placebo Then Guanfacine
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: Second Intervention (Day 4)
Arm/Group | Guanfacine Then Placebo | Placebo Then Guanfacine
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Drug and Placebo: All patients will receive a single dose of drug and a single dose of placebo on separate days of the trial period. The order in which they receive these will be randomized.
  Guanfacine: 2mg oral guanfacine (encapsulated)
  Placebo: placebo
Arm/Group | Drug and Placebo
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 13
Behavioural Inattention Test Star Cancellation Score (Total targets found) [Mean (Standard Deviation); unit: Number of targets found] — This is a standard scale for measuring the severity of spatial neglect. Patients are asked to find and mark targets (which are embedded amongst distractors) on a piece of paper. The maximum number of targets that can be found is 54 (Therefore minimum score =0, maximum =54), which represents normal performance.
  Number of targets found | 35.4 (15.9)
Mesulam Shape Cancellation Score (Total targets found) [Mean (Standard Deviation); unit: Number of targets found] — This is a standard scale for measuring the severity of spatial neglect. Patients are asked to find and mark targets (which are embedded amongst distractors) on a piece of paper. The maximum number of targets that can be found is 60 (Therefore minimum score =0, maximum = 60), which represents normal performance.
  Number of targets found | 25.6 (13.7)
Touchscreen Cancellation [Mean (Standard Deviation); unit: Number of targets found] — This is a computerised scale for measuring the severity of spatial neglect as described in previous publications (Malhotra et al, Annals of Neurology 2006; Parton et al, Neuroreport 2006). Patients are asked to find and touch targets (which are embedded amongst distractors) on a touchscreen. In the variant of the task employed here, the targets are not marked when touched ("Invisible Cancellation").The maximum number of targets that can be found is 64 (Therefore minimum score = 0, maximum = 64), which represents normal performance.
  Number of targets found | 28.4 (13.9)

OUTCOME MEASURES:

1. Primary Outcome: Performance on Tests of Hemispatial Neglect and Sustained Attention
Description: Touchscreen Cancellation: This is a computerised scale for measuring the severity of spatial neglect as described in previous publications (Malhotra et al, Annals of Neurology 2006; Parton et al, Neuroreport 2006). Patients are asked to find and touch targets (which are embedded amongst distractors) on a touchscreen. In the variant of the task employed here, the targets are not marked when touched ("Invisible Cancellation").The maximum number of targets that can be found is 64 (Therefore minimum score =0, maximum = 64), which represents normal performance.
Time Frame: 5 days
Population: Baseline performance was determined for each patient by averaging scores on days 1, 3 and 5, as well as the preadministration sessions on days 2 and 4. Group averages and differences were computed between treatment type (baseline, guanfacine and placebo) across individuals.
Measure: Mean (Standard Deviation); unit: Number of targets found
Groups:
- All Patients: All individuals received guanfacine and placebo in a crossover design.
Arm/Group | All Patients
Number analyzed (Participants) | 13
Number of targets found
  Touchscreen Cancellation-Guanfacine | 31.15 (15.1)
  Touchscreen Cancellation-Placebo | 26.15 (14.29)
Statistical Analysis 1: Comparison: All Patients; between the placebo and guanfacine conditions; Test type: Superiority; p = 0.013, t-test, 2 sided

2. Secondary Outcome: Performance on Motor Tasks
Description: Time taken to take pegs from a container and place them into holes on a board, and then remove these pegs and replace them in the container.
Time Frame: 5 Days
Population: All patients were unable to carry out this task (9 hold PEG test of finger dexterity) because of the paralysis caused by their stroke.
Groups:
- All Patients: All patients received guanfacine then placebo or vice versa.
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

LIMITATIONS AND CAVEATS:
The trial involved a single dose of active drug and a single dose of placebo given in a crossover design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes